CLINICAL TRIAL: NCT06573177
Title: Gender Incongruence in Danish Youth (GenDa): An Observational Cohort Study of Danish Children and Adolescents Referred to a National Gender Identity Service
Brief Title: Optimizing Individual Health Care for Young People With Gender Incongruence
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Katharina Maria Main, Prof. MD, Ph.d., Rigshospitalet, Denmark
Other Study IDs: H-18050607
Record Dates: First submitted 2024-04-18; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Gender Incongruence
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, plasma, DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Referral to the gender identity service. — Referral to the national gender identity service consisting of the Sexological Clinic, Child and Adolescent Mental Health Center, and Department of Growth and Reproduction in the Capital Region of Denmark.

SUMMARY:
This observational study focuses on evaluating the effect of the current health care program for Danish children and adolescents with gender incongruence, which was established in January 2016. Somatic outcome parameters include growth, bone health, body composition, metabolic parameters, hormone levels and concurrent diseases. Psychosocial parameters include the trajectory of gender incongruence development, mental health, i.e. autism spectrum disorders, behavioural problems, self-harm, suicidal ideation and psychiatric diagnoses, and social context, i.e. family demographics, education, minority stress.

This study aims to:

1. Characterise the psychosocial profile of all children and adolescents referred for treatment, as well as the history of gender identity development and treatment trajectories.
2. Systematically evaluate biological parameters before and during hormonal treatment with gonadotropin-releasing hormone (GnRH) analogues and cross-sex hormones, and to establish a biobank for those in hormone treatment.

The investigators hypothesise that intervention with counselling and hormonal treatment is safe and has a positive impact on psychosocial well-being of transgender youngsters. The overall aim is to provide data for improving future family counselling, clinical care, patient satisfaction, patient safety and ultimately quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* Accepted referral to the gender identity service.

Exclusion Criteria:

* None.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children and youngsters under the age of 18 years referred to the gender identity service in Denmark.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 8 years
  BMI will be calculated from height and weight (kg/m^2) measurements
Puberty | 8 years
  Tanner stages of puberty (1-5) are obtained by clinical examination
Bone mineral content (BMD) | 8 years
  Whole body dual-energy x-ray absorptiometry (DXA) will determine BMD Z-score for age and sex
Body fat | 8 years
  Whole body dual-energy x-ray absorptiometry (DXA) will measure body fat percentage (%)
Lean body mass | 8 years
  Whole body dual-energy x-ray absorptiometry (DXA) will measure lean mass (kg)
Reproductive serum hormone levels | 8 years
  Changes in reproductive hormone levels (%)
Adrenal serum hormone levels | 8 years
  Changes in adrenal hormone levels (%)
Blood pressure | 8 years
  Changes in blood pressure measurement (mm Hg)
Transabdominal ultrasound of uterus | 8 years
  Changes of endometrium (thickness in mm) during testosterone treatment
Transabdominal ultrasound of ovaries | 8 years
  Change in number of follicles (n) during testosterone treatment
Sperm count | 8 years
  Sperm Count (at cryopreservation)
Sperm motility | 8 years
  Sperm motility (at cryopreservation)
Morbidity | 8 years
  Number of participants with registered ICD10 diagnoses
Demographic characteristics | 8 years
  eg. socioeconomic status
Prevalence of psychiatric disorders | 8 years
  Based on screening for psychopathology using validated tests, as indicated:
  Schedule for Affective Disorders and Schizophrenia for School-age children (K-SADS):
  A diagnostic tool used to assess psychiatric disorders in children and adolescents. It is a semi-structured interview guide used to identify psychiatric conditions.
  Wechsler Intelligence Scale for Children (WISC 4/5) or Wechsler Adult Intelligence Scale (WAIS 4): General cognitive function is measured on a scale from 40-160 which is used as an intelligence quotient. A higher score: A higher cognitive function.
  Rorschach: A projective psychological test. The test uses a series of ink blots to evaluate a person's mental functions and emotional state by analysing their perceptions of the figures. The test is based on complex and subjective scoring and interpretation.
Prevalence of Attention Deficit Hyperactive Disorder (ADHD) | 8 years
  Screening using validated tests:
  Behavior Rating Inventory of Executive Function (BRIEF): General executive function is measured on a normative scale with T-scores from 20-80. A higher score: more executive difficulties.
  Attention Deficit/Hyperactive Disorder-Rating Scale (ADHD-RS): Attention Deficit Hyperactive Disorder traits measured on a normative scale with T-scores from 0-78. A higher score: More Attention Deficit Hyperactive Disorder traits
Prevalence of autism spectrum disorder | 8 years
  Screening using validated tests:
  Social Responsiveness Scale (SRS): Autism spectrum disorder (ASD) traits measured on a scale with T-scores from 0-76+. A higher score: More autistic traits.
  Autism Diagnostic Observation Schedule (ADOS): A structured observational tool to assess ASD. A trait is rated on a scale from 0 to 3. 0 indicates absence of a behaviour and 3 indicates severe occurrence of a behaviour. The total score determines the presence and severity of ASD. The cut-off scores are 10 for autism and 7 for ASD traits.
  Autism Diagnostic Interview-Revised (ADI-R): A structured interview used to assess ASD traits. Interview questions are scored on a scale from 0-3. 0 indicates absence of a behaviour and 3 indicates severe occurrence of a behaviour. The scores compared with cut-off values determine the presence of ASD. Cut-off values for each trait: Social interaction: cut-off 10; Communication skills: cut-off 8; Restrictive and repetitive behaviour patterns: cut-off 3.
Global level of functioning | 8 years
  Children's Global Assessment Scale (C-GAS, range 1-100)
Psychosocial Disability | 8 years
  Global Assessment of Psychosocial Disability (GAPD, range 0-8)
Suicide risk | 8 years
  Number of participants with self-reported suicide thoughts or attempts (interview)
Substance abuse. | 8 years
  Number participants with self-reported abuse of alcohol, drugs or medications (interview)
Personal history of gender incongruence (GI) | 8 years
  Age at onset of GI and social transitioning (interview)
Cultural measures | 8 years
  Interviews with youngsters and their families to explore:
  1) The experiences that are influential in the process of seeking gender-affirming treatment. 2) Treatment expectations and wishes. 3) The cultural understandings of gender, sex, body and identity that inform the decision to seek treatment. 4) The role of the family in the decision to seek treatment.
Establishment of biobank | 8 years.
  Serum, plasma, DNA at -20 and -80 degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina M Main, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No